CLINICAL TRIAL: NCT00569738
Title: Ga68-DOTA-NOC-PET Imaging of Neuroendocrine Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Yodphat Krausz M.D., Hadassah Medical Organization
Other Study IDs: 061267-HMO-CTIL; Imaging of NE Tumors
Record Dates: First submitted 2007-12-06; First posted 2007-12-07 (Estimated); Last update posted 2009-02-17 (Estimated); Status verified 2009-02

CONDITIONS: Neuroendocrine Tumor
Keywords: neuroendocrine tumor; somatostatin analog; Gallium 68; PET
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: patients with neuroendocrine tumors
  Interventions: Procedure: PET scan with Ga68-DOTANOC

INTERVENTIONS:
Procedure: PET scan with Ga68-DOTANOC — Imaging: PET scan with Ga68-DOTANOC

SUMMARY:
Imaging of neuroendocrine tumors (NETs) relies on conventional morphological methods and on somatostatin receptor scintigraphy (SRS). SRS is effective for carcinoid tumors, and for most pancreatic islet-cell tumors, but may fail to detect some tumors. Furthermore, this technique may require repeated imaging over 24-48 hours. Introduction of newer somatostatin analogs such as DOTANOC improves lesion detection. In addition, labeling with Ga68 and use of PET/CT improves the pharmacokinetics of the tracer resulting in better tumor visualization, and an easier procedure with imaging over only 1-2 hours.

In this study, we propose to use Ga68-DOTANOC PET for imaging of various NETs, comparing the imaging data to those of anatomical and other functional modalities, and to histopathology, when available.

DETAILED DESCRIPTION:
Neuroendocrine tumors (NETs), best treated by complete surgical resection, are frequently difficult to localize due to small size, presence in hollow organs, and morphological changes caused by prior surgery. Imaging of NETs relies primarily on conventional morphological methods (EUS, CT, MRI, US). Functional imaging, such as somatostatin receptor scintigraphy (SRS) using the In111-labeled somatostatin analog octreotide, provides better staging of the disease, visualization of occult tumor, and evaluation of patient eligibility for somatostatin analog treatment. This modality is effective for carcinoid tumors, and for most pancreatic islet-cell tumors. However, it may fail to detect some tumors, mostly due to low density of somatostatin receptors, with resulting lack of tumor uptake. The relatively poor spatial resolution of planar and SPECT imaging may also reduce tumor detection, particularly for small tumors and/or those with low uptake. Furthermore, this technique is lengthy, often requiring repeated imaging over 24-48 hours. Introduction of newer somatostatin analogs such as DOTANOC offers many advantages. Higher uptake of the newer analogs in more of the somatostatin receptor subtypes improves lesion detection. In addition, labeling with the positron emitter, Ga68, instead of In111 improves the pharmacokinetics of the tracer, and the faster tumor uptake and more rapid clearance from normal tissues increases tumor to background contrast, improving tumor visualization, and resulting in an easier procedure with imaging only 1-2 hours after tracer injection. The superior spatial resolution of positron emission tomography (PET) again enhances lesion detectability, and use of PET makes it possible to perform exact quantitation of tracer uptake that can be useful for monitoring therapy and for planning peptide receptor radionuclide therapy.

In this study, we propose to use Ga68-DOTANOC PET for imaging of various NETs, comparing the imaging data to those of anatomical and other functional modalities, and to histopathology, when available.

ELIGIBILITY:
Inclusion Criteria:

* neuroendocrine tumor
* patients who are able to lie in scanner for up to 50 minutes

Exclusion Criteria:

* under age 18
* pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: neuroendocrine tumor clinic
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2008-12; Study Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yodphat Krausz, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Department of Nuclear Medicine, Hadassah Medical Center, Jerusalem, Israel